CLINICAL TRIAL: NCT05218330
Title: Weekend Headaches in School-age Children
Brief Title: The Incidents of Weekend Headaches in Children
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Principal Investigator, Jacob.genizi, Director Pediatric Departement, Bnai Zion Medical Center
Other Study IDs: bnz 0138-21
Record Dates: First submitted 2022-01-27; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Headache; Child, Only
Keywords: HEADACHE; CHILDREN; WEEKENDS
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational prospective follow-up study. The study population will include 30 children aged 6-18 years who suffer from a primary headache and are treated at the Pediatric Neurology Clinic at Bnai Zion Hospital in Haifa, Israel.

After the adolescents or parents sign an informed consent to participate in the study, they will receive a headache diary (Appendix 1) which they will fill out for 4 weeks as recommended [15]. They will mark the day the headache appeared, its intensity, duration, and timing during the day. In addition, they will fill the various triggers offered (such as sleep hours, exercise time, screen hours, and a subjective sense of academic or emotional stress) on days with headache and on every weekend.

We will then divide the participants into two groups - those who suffer from a headache in the middle of the week only (MWH) and those who suffer from a headache at the weekend (WH), compare the demographic and clinical characteristics and we will try to understand the triggers of these two groups.

Patients will also be asked a questionnaire which will define whether they are having difficulty in school (Appendix 2) so that we can examine the distribution of headaches of this group during the week.

A physician who works on the research team will proactively verify that the questionnaire is filled out consistently and accurately. Additional data will be collected from the medical record.

DETAILED DESCRIPTION:
Research topic:

Weekend headaches in school-age children

Scientific background:

Headache is one of the most common complaints in children and adolescents. It is recognized as one of the top medical and neurologic contributors to the global burden of disease and is a leading cause of disability in adolescents and young adults [1].

Recurrent severe headaches also are common in children. In the United States, approximately 20 percent of children aged 4 to 18 years report having had notable recurrent headaches in the past 12 months and the prevalence increases with age [2].

The International Classification of Headache Disorders, 3rd edition (ICHD-3) provides detailed diagnostic criteria for primary headaches which include mainly migraine and tension-type headache [3].

A diary in which the quality, location, severity, timing, precipitating and palliating factors, and associated features of the headache are recorded prospectively (not subject to recall error) may be a useful adjunct if the child is willing and able to complete daily [4].

There are many triggers for headaches including academic or emotional stress, lack of sleep, or lack of exercise, multiple screen hours, untidy meals, change in consumption of caffein, alcohol or energy drinks, etc. It can be assumed that the presence of these triggers varies between weekends and routine days at school and thus affects the incidence of headache [5-8].

There are few studies that investigated weekend headaches among the adult population [9-11], and only two studies which mentioned differences in headache between days of the week among school [12, 13]. Mehta [12] reported the rate of headaches in weekends to be 5.9% compared to 28.5% on monday, among children age 7-14 years of age. However they didn't report on the incidence of other weekdays headaches. On the other hand, Larsson et al [13] didn't find significant difference in headache incidence between weekdays and weekends, although the peak incidence was at the middle of at Thursday.

Finally, learning disabilities and ADHD are more common in children and adolescents who suffer from primary headaches [14], and because much of the headache in children is attributed to school, it will be interesting to see the effect of this group on the distribution of headache throughout the week.

Purpose of the study:

Our goal is to investigate whether there is weekend headache in children and adolescents and what are the risk factors.

Methods:

This is an observational prospective follow-up study. The study population will include 30 children aged 6-18 years who suffer from a primary headache and are treated at the Pediatric Neurology Clinic at Bnai Zion Hospital in Haifa, Israel.

After the adolescents or parents sign an informed consent to participate in the study, they will receive a headache diary (Appendix 1) which they will fill out for 4 weeks as recommended [15]. They will mark the day the headache appeared, its intensity, duration, and timing during the day. In addition, they will fill the various triggers offered (such as sleep hours, exercise time, screen hours, and a subjective sense of academic or emotional stress) on days with headache and on every weekend.

We will then divide the participants into two groups - those who suffer from a headache in the middle of the week only (MWH) and those who suffer from a headache at the weekend (WH), compare the demographic and clinical characteristics and we will try to understand the triggers of these two groups.

Patients will also be asked a questionnaire which will define whether they are having difficulty in school (Appendix 2) so that we can examine the distribution of headaches of this group during the week.

A physician who works on the research team will proactively verify that the questionnaire is filled out consistently and accurately. Additional data will be collected from the medical record.

The study will be conducted after receiving approval from the Institutional Helsinki Committee

Statistical analysis:

The data will be processed and analyzed using SPSS software. Two sample t-test will be performed for continuous variables, and X² for categorial data. Odds ratios with 95% confidence intervals will be computed, statistical significance is considered as p <0.05.

Tables and graphs:

Appendix 1- Headache diary (לצרף Appendix 2- Questionnaire to diagnose suspected difficulty in studies (לצרף? Table 1- Demographic characteristics of children with weekend headache and children without weekend headache Weekend headache (WH) Midweek headache (MWH) P value Number of children, no. (%) 10 (33) 20 (67) Age, years, mean Sex, % Boys Girls Ethnicity, % Jewish Arab Other

Table 2- Clinical characteristics of children with weekend headache and children without weekend headache Weekend headache (WH) Midweek headache (MWH) P value Severity, mean Duration, hours, mean Timing during the day (morning/evening) Type of headache Migraine Tension type headache Mixed Other learning disabilities % Other somatic complaints %

Table 3- Lifestyle and stress triggers over the weekend Weekend headache (WH) Midweek headache (MWH) P value Academic stress (1-5), mean Emotional stress (1-5), mean Hours of sleep at night, mean Sportive activity (1-5), mean Regular meals (1-5), mean Screen hours, mean

ELIGIBILITY:
Inclusion Criteria:

* Children age 6-18 years old with primary headaches
* Attending school

Exclusion Criteria:

* Secondary headaches
* Developmental delay
* Malignancy

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children age 6-18 years old with normal development attending scool
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
weekends headaches frequency | 1 year
  Are weekdays headaches frequent in school children more than in weekends? We will use a pen headache diary to asses headache frequency

SECONDARY OUTCOMES:
weekends headaches frequency risk factors | 1 year
  To investigate the risk factors for pediatric weekends headaches. We will use a questionnaire to asses sleeping hours, sport, meals and other triggers.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob genizi, md, Principal Investigator — Bnai Zion Medical Center
Locations (1):
- Bani Zion, Haifa, Israel

REFERENCES:
- [Result] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Result] Lateef TM, Merikangas KR, He J, Kalaydjian A, Khoromi S, Knight E, Nelson KB. Headache in a national sample of American children: prevalence and comorbidity. J Child Neurol. 2009 May;24(5):536-43. doi: 10.1177/0883073808327831. PMID 19406755
- [Result] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Result] van den Brink M, Bandell-Hoekstra EN, Abu-Saad HH. The occurrence of recall bias in pediatric headache: a comparison of questionnaire and diary data. Headache. 2001 Jan;41(1):11-20. doi: 10.1046/j.1526-4610.2001.111006011.x. PMID 11168599
- [Result] Gariepy G, Dore I, Whitehead RD, Elgar FJ. More than just sleeping in: a late timing of sleep is associated with health problems and unhealthy behaviours in adolescents. Sleep Med. 2019 Apr;56:66-72. doi: 10.1016/j.sleep.2018.10.029. Epub 2018 Nov 20. PMID 30545801
- [Result] Rogers DG, Bond DS, Bentley JP, Smitherman TA. Objectively Measured Physical Activity in Migraine as a Function of Headache Activity. Headache. 2020 Oct;60(9):1930-1938. doi: 10.1111/head.13921. Epub 2020 Aug 2. PMID 32740940
- [Result] Toyran M, Ozmert E, Yurdakok K. Television viewing and its effect on physical health of schoolage children. Turk J Pediatr. 2002 Jul-Sep;44(3):194-203. PMID 12405429
- [Result] Couturier EG, Hering R, Steiner TJ. Weekend attacks in migraine patients: caused by caffeine withdrawal? Cephalalgia. 1992 Apr;12(2):99-100. doi: 10.1046/j.1468-2982.1992.1202099.x. PMID 1576651
- [Result] Drescher J, Wogenstein F, Gaul C, Kropp P, Reinel D, Siebenhaar Y, Scheidt J. Distribution of migraine attacks over the days of the week: Preliminary results from a web-based questionnaire. Acta Neurol Scand. 2019 Apr;139(4):340-345. doi: 10.1111/ane.13065. Epub 2019 Jan 28. PMID 30636039
- [Result] Torelli P, Cologno D, Manzoni GC. Weekend headache: a retrospective study in migraine without aura and episodic tension-type headache. Headache. 1999 Jan;39(1):11-20. doi: 10.1046/j.1526-4610.1999.3901011.x. PMID 15613189
- [Result] Torelli P, Cologno D, Manzoni GC. Weekend headache: a possible role of work and life-style. Headache. 1999 Jun;39(6):398-408. doi: 10.1046/j.1526-4610.1999.3906398.x. PMID 11279917
- [Result] Mehta S. Study of various social and demographic variables associated with primary headache disorders in 500 school-going children of central India. J Pediatr Neurosci. 2015 Jan-Mar;10(1):13-7. doi: 10.4103/1817-1745.154319. PMID 25878735
- [Result] Larsson B, Fichtel A. Headache prevalence and characteristics among school children as assessed by prospective paper diary recordings. J Headache Pain. 2012 Mar;13(2):129-36. doi: 10.1007/s10194-011-0410-9. Epub 2011 Dec 27. PMID 22200765
- [Result] Genizi J, Gordon S, Kerem NC, Srugo I, Shahar E, Ravid S. Primary headaches, attention deficit disorder and learning disabilities in children and adolescents. J Headache Pain. 2013 Jun 27;14(1):54. doi: 10.1186/1129-2377-14-54. PMID 23806023
- [Result] Osterhaus SO, Passchier J. The optimal length of headache recording in juvenile migraine patients. Cephalalgia. 1992 Oct;12(5):297-9. doi: 10.1046/j.1468-2982.1992.1205297.x. PMID 1423561